CLINICAL TRIAL: NCT02052869
Title: Spirometric Detection of Esophageal Intubation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has left the hopsital
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Lazarus 003
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Hypoxia; Hypoventilation
Keywords: endotracheal intubation; esophageal intubation
MeSH Terms: conditions — Hypoxia; Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- esophagus intubation (Other): all patients will be intubated in the trachea first, with subsequent intubation in the esophagus. measurements will be performed on both tubes in a blinded manner.
  Interventions: Procedure: esophagus intubation

INTERVENTIONS:
Procedure: esophagus intubation — In these patients, automatic pressure waveform analysis is performed during the first three test ventilations on both the tracheal and oesophageal tube. ventilations will be performed by a blinded person. Subsequently, three conventional thoracic pushes will be performed.

SUMMARY:
In endotracheal intubation, it is essential that the trachea is intubated and not the esophagus. In suboptimal situations (outside an operating theatre), malpositioning of the endotracheal tube occurs frequently and is often fatal. The diagnostic tools that are available in the operating theatre are not appropriate for out-of-hospital situations because of several reasons. Moreover, these methods mostly take some time to provide the desired information and don't have optimal specificity and sensitivity. In order to allow fast diagnosis of this potentially fatal complication, we have developed a fully-automatic detection device to diagnose endotracheal tube malpositioning within 2 seconds.

A high sensitivity/specificity of the algorithm for waveform-analysis was demonstrated in healthy patients and patients with pulmonary diseases (decreased pulmonary compliance).

A new stand-alone device with integrated sensors and microprocessor was developed that gives immediate diagnosis, and stores data for subsequent research purpose. This device will be evaluated in perioperative situations to demonstrate the high sensitivity and specificity in patients in a clinical setting.

DETAILED DESCRIPTION:
The fundamental algorithm for waveform analysis is unchanged, but an additional detection algorithm is incorporated for improved detection of ventilation efforts. In addition, sensors are integrated, automatic feedback electronics are improved, and the device is made more user friendly to be appropriate for out-of-hospital situations in demanding environments.

In addition, waveforms will be recorded for later analysis and evaluation of the diagnostic value of a thoracic push ( a gentle push on the sternum) to detect tube position.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia with endotracheal intubation required for the procedure
* Age: 18 years and older
* Total intravenous anesthesia with propofol (in order ro guarantee adequate hypnosis during the procedure)

Exclusion Criteria:

* Oesophageal pathology
* Patients at risk for desaturation (SpO2 < 95%) if 20 seconds of apnoea is induced after adequate preoxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
sensitivity/specificity of the fully-automatic device | first 3 minutes after intubation
  Determine the sensitivity/specificity of the fully-automatic device to diagnose oesophageal intubation based on test ventilations

SECONDARY OUTCOMES:
Evaluate the value of the supplementary algorithm | first 3 minutes of intubation
  Evaluate the value of the supplementary algorithm to detect tube position without test ventilation. relying on only pressure waveform analysis during a conventional "thoracic push"

CONTACTS AND LOCATIONS:
Overall Officials: Alain Kalmar, MD PhD, Principal Investigator — University hosptal Medical Center Groningen,University of Groningen, The Netherlands
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands